CLINICAL TRIAL: NCT00066872
Title: A Randomized Controlled Trial of Excisional Surgery Versus Imiquimod 5% Cream for Nodular and Superficial Basal Cell Carcinoma
Brief Title: Topical Imiquimod Compared With Surgery in Treating Patients With Basal Cell Skin Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000320513; CRUK-LON-SINS-C7484/A2869; EU-20205
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Imiquimod

INTERVENTIONS:
Drug: imiquimod
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies such as imiquimod use different ways to stimulate the immune system and stop cancer cells from growing. It is not yet known if topical imiquimod is more effective than surgery in treating basal cell skin cancer.

PURPOSE: This randomized phase III trial is studying how well topical imiquimod works compared to surgery in treating patients with basal cell skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the rate of local recurrence at 3 years in patients with nodular or superficial basal cell skin cancer treated with imiquimod 5% cream vs excisional surgery.
* Compare recurrence at 6 months and 1, 2, and 5 years in patients treated with these regimens.
* Compare the time to first recurrence in patients treated with these regimens.
* Compare the aesthetic appearance of lesion sites in patients treated with these regimens.
* Compare pain in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and lesion type (nodular vs superficial). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive topical imiquimod to a single lesion once daily for 6 weeks for a superficial lesion or 12 weeks for a nodular lesion. Patients with early treatment failure or recurrence are offered surgical excision.
* Arm II: Patients undergo surgical excision. Patients are followed at 6, 12, and 18 weeks, every 6 months for 1 year, annually for 2 years, and then at 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary basal cell skin carcinoma

  * Nodular or superficial lesion(s)*
  * Located in low-risk areas NOTE: *Any number of lesions are allowed but only 1 lesion per patient is selected for the study
* No genetic or nevoid conditions (e.g., Gorlin's syndrome)
* No morphoeic (microinfiltrative) histology

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No bleeding disorder

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 1 month after study participation
* No allergy to any of the study interventions
* No life-threatening disease
* Must be available for study follow-up for up to 3 years
* Must have access to a telephone

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent participation in any other experimental trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2002-10; Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Absence of local recurrence at 3 years after start of treatment

SECONDARY OUTCOMES:
Recurrence of basal cell cancer (BCC) at 1, 2, and 5 years
Time to first occurrence up to 5 years from completion of study treatment
Aesthetic appearance of lesion site as measured by participant and blind observer using 5-point Likert scale at 6 months, and then years 1-3
Pain at lesion site as measured by 6-point scale daily during treatment, and then 16 weeks after the completion of study treatment
Cost effectiveness assessed up to 3 or 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mara Ozolins, MS — Queen's Medical Center
Locations (3):
- United Kingdom (3):
  - Chesterfield Royal Hospital, Chesterfield, England
  - Queen's Medical Centre, Nottingham, England
  - Solihull Hospital, Solihull, England

REFERENCES:
- [Result] Ozolins M, Williams HC, Armstrong SJ, Bath-Hextall FJ. The SINS trial: a randomised controlled trial of excisional surgery versus imiquimod 5% cream for nodular and superficial basal cell carcinoma. Trials. 2010 Apr 21;11:42. doi: 10.1186/1745-6215-11-42. PMID 20409337
- [Derived] Williams HC, Bath-Hextall F, Ozolins M, Armstrong SJ, Colver GB, Perkins W, Miller PSJ; Surgery Versus Imiquimod for Nodular and Superficial Basal Cell Carcinoma (SINS) Study Group. Surgery Versus 5% Imiquimod for Nodular and Superficial Basal Cell Carcinoma: 5-Year Results of the SINS Randomized Controlled Trial. J Invest Dermatol. 2017 Mar;137(3):614-619. doi: 10.1016/j.jid.2016.10.019. Epub 2016 Dec 5. PMID 27932240
- [Derived] Bath-Hextall F, Ozolins M, Armstrong SJ, Colver GB, Perkins W, Miller PS, Williams HC; Surgery versus Imiquimod for Nodular Superficial basal cell carcinoma (SINS) study group. Surgical excision versus imiquimod 5% cream for nodular and superficial basal-cell carcinoma (SINS): a multicentre, non-inferiority, randomised controlled trial. Lancet Oncol. 2014 Jan;15(1):96-105. doi: 10.1016/S1470-2045(13)70530-8. Epub 2013 Dec 11. PMID 24332516